CLINICAL TRIAL: NCT04756713
Title: Impact of Second Uterine Evacuation in Women With Non-metastatic, Low-risk Gestational Trophoblastic Neoplasia: A Phase III Trial
Brief Title: Second Uterine Evacuation for Low-risk Gestational Trophoblastic Neoplasia
Acronym: ReCure
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Maternidade Escola da Universidade Federal do Rio de Janeiro (Unknown); Universidade Federal do Rio de Janeiro (Other); Federal University of Ceará (Unknown); Federal University of São Paulo UNIFESP (Unknown); Campinas State University UNICAMP (Unknown); Paulista State University UNESP BOTUCATU (Unknown); Medical School of Santa Casa da Misericórdia de Porto Alegr (Unknown); University of Caxias do Sul (Unknown)
Responsible Party: Principal Investigator, Kevin Elias, Co-investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ReCure
Record Dates: First submitted 2021-02-12; First posted 2021-02-16 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Gestational Trophoblastic Neoplasia; Molar Pregnancy; Gestational Trophoblastic Tumor, Non-Metastatic
MeSH Terms: conditions — Gestational Trophoblastic Disease; Hydatidiform Mole | interventions — Vacuum Curettage; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Investigator, Outcomes Assessor
Masking Description: Treatment assignments are made by a remote investigator not involved in the clinical care of the patient using a coded key with random block sizes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy (Active Comparator): Patients allocated to receive conventional chemotherapy will be treated with methotrexate (1 mg/kg intramuscular) with rescue of folinic acid (15mg orally). In cases of chemoresistance, second-line chemotherapy will be performed with actinomycin-D (Act-D) 1.25 mg intravenous pulse every 14 days. The third line of chemotherapy will be the EMA/CO regimen (reserving the EP / EMA regimen (E, cisplatin, MTX / Act-D) for the fourth line.
  Interventions: Drug: Chemotherapy
- Uterine evacuation (Experimental): Patients randomized to undergo a second curettage will undergo manual or electronic vacuum aspiration under ultrasound guidance. Following discharge after the second curettage patients will return to weekly hCG monitoring. If hCG levels are decreasing, patients will remain on weekly hCG follow-up until the first normal hCG (<5 IU/L) is achieved. Then they will have monthly hCG monitoring for 12 months. If patients do not attain remission and develop persistent GTN as established by FIGO 2000, the tumor will be re-staged and appropriate chemotherapy will be initiated.
  Interventions: Procedure: Uterine curettage

INTERVENTIONS:
Procedure: Uterine curettage — Manual or electric vacuum aspiration under ultrasound guidance.
  Arms: Uterine evacuation
Drug: Chemotherapy — conventional chemotherapy will be treated with MTX (1 mg/kg intramuscular) with rescue of FA (15mg orally). In cases of chemoresistance, second-line chemotherapy will be performed with actinomycin-D (Act-D) 1.25 mg intravenous pulse every 14 days. The third line of chemotherapy will be the EMA/CO regimen (, reserving the EP / EMA regimen (E, cisplatin, MTX / Act-D) for the fourth line.
  Arms: Chemotherapy

SUMMARY:
To evaluate the efficacy and safety of second uterine curettage in patients with low-risk non-metastatic GTN.

DETAILED DESCRIPTION:
This is a randomized, multicenter clinical trial including patients seen at one of 13 gestational trophoblastic disease reference centers in Brazil. Subjects are eligible if they have low-risk gestational trophoblastic neoplasia according to FIGO 2000 criteria and the FIGO/WHO prognostic risk score. The study includes two treatment arms: immediate treatment with single-agent chemotherapy (center choice of agent) or second uterine curettage. The primary outcome is the rate of primary remission. Secondary outcomes are the number of chemotherapy cycles required to achieve remission, rate of primary chemotherapy resistance, rate of relapse, and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of molar pegnancy according to the morphological criteria described by Sebire et al., who meet the diagnostic criteria for low-risk non-metastatic GTN according to FIGO 2000 criteria

Exclusion Criteria:

1. High risk GTN (FIGO risk score ≥ 7) or metastatic disease at diagnosis of GTN (stage II, III or IV);
2. Histopathological diagnosis of choriocarcinoma, placental site trophoblastic or epithelioid trophoblastic tumor at the second curettage;
3. Previous chemotherapy treatment;
4. Level of hCG at the time of GTN diagnosis less than 20 IU/L (to minimize the risk of inclusion of patients with false positive hCG, either by cross-reaction with pituitary hormones or by the presence of circulating heterophilic antibodies);
5. Relapsed GTN;
6. Incomplete medical records.
7. Loss to follow-up;
8. Voluntary desire to stop participating in the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-02-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Remission rate from primary therapy | 3 years
  Undetectable hCG on weekly serum assay for at least three weeks

SECONDARY OUTCOMES:
Cycles to remission | 3 years
  Total number of cycles of chemotherapy required to attain remission
Time to remission | 3 years
  Time in days from randomization to remission
Need for multiagent chemotherapy | 3 years
  Need for progression from single agent to multiagent chemotherapy
Relapse | 1 year
  Re-elevation of hCG after achieving remission
Death | 1 year
  Death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Braga, MD, PhD, Study Director — Maternidade Escola da Universidade Federal do Rio de Janeiro
Locations (7):
- Brazil (7):
  - Paulista State University UNESP, Botucatu
  - Campinas State University UNICAMP, Campinas
  - University of Caxias do Sul, Caxias do Sul
  - Federal University of Ceará, Ceará
  - Medical School of Santa Casa da Misericórdia de Porto Alegre, Porto Alegre
  - Maternidade Escola da Universidade Federal do Rio de Janeiro, Rio de Janeiro
  - Federal University of São Paulo UNIFESP, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Osborne RJ, Filiaci VL, Schink JC, Mannel RS, Behbakht K, Hoffman JS, Spirtos NM, Chan JK, Tidy JA, Miller DS. Second Curettage for Low-Risk Nonmetastatic Gestational Trophoblastic Neoplasia. Obstet Gynecol. 2016 Sep;128(3):535-542. doi: 10.1097/AOG.0000000000001554. PMID 27500329
- [Background] Hemida R, Vos EL, El-Deek B, Arafa M, Toson E, Burger CW, van Doorn HC. Second Uterine Curettage and the Number of Chemotherapy Courses in Postmolar Gestational Trophoblastic Neoplasia: A Randomized Controlled Trial. Obstet Gynecol. 2019 May;133(5):1024-1031. doi: 10.1097/AOG.0000000000003232. PMID 30969220